CLINICAL TRIAL: NCT04888104
Title: Prospective, Multicenter, Case-Control Analysis of the VersaTie Posterior Fixation System to Prevent Proximal Junctional Failure in Long Posterior Spinal Fusion Constructs for Adult Patients
Status: Recruiting | Type: Observational
Sponsor: International Spine Study Group Foundation (Other)
Collaborators: NuVasive (Industry)
Responsible Party: Sponsor
Other Study IDs: 2139
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Adult Spinal Deformity; Scoliosis; Kyphosis
Keywords: Scoliosis; Kyphosis; Sagittal Imbalance
MeSH Terms: conditions — Scoliosis; Kyphosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Procedure: Index or revision spine surgery for complex adult spinal deformity — Adult patients receiving minimum 5 level posterior spinal fusion with pedicle screw fixation supplemented at the proximal aspect of the construct with the VersaTie System.
  Other Names: VersaTie System

SUMMARY:
Prospective, Multicenter, Case-Control Analysis of the VersaTie Posterior Fixation System to Prevent Proximal Junctional Failure in Long Posterior Spinal Fusion Constructs for Adult Patients

DETAILED DESCRIPTION:
Specific Aims:

* Evaluate the safety and performance of posterior spinal fusion constructs supplemented with posterior spinolaminar fixation using the VersaTie System compared to posterior fixation constructs without VersaTie System supplementation in adult patients undergoing long posterior spinal fusion by evaluating intraoperative and postoperative complications, clinical and radiographic outcomes, patient-reported outcomes (PROs) and need for revision surgery.
* Evaluate surgical treatment outcomes and identify best practice guidelines for complex adult spinal deformity (ASD) patients, including radiographic and clinical outcomes, surgical and postoperative complications, risk factors for and revision surgery.
* Develop and validate a standardized, universal complications classification system for spine surgery
* Evaluate perioperative blood management approaches, transfusion requirements, including variance in thresholds for blood transfusion and associated complications for adult spinal deformity surgery
* Assess impact of opioid use and pain management on patient cost, complications and outcomes
* Evaluate optimal opioid and analgesic usage and protocols for standard work development
* Evaluate clinical outcomes utilizing legacy patient reported outcome measures (PROMs) including modified Oswestry Disability Index (mODI), Scoliosis Research Society Questionnaire 22r (SRS-22r), Veterans RAND-12 (VR-12), and numeric pain rating scale (NRS) and compare the results of these legacy PROMs to outcomes scores as measured by the NIH Patient Reported Outcomes Measurement Information System (PROMIS) - PROMIS Anxiety, Depression, Pain Interference, Physical Function, and Social Satisfaction. Secondary aims for PROM research for this study include

  1. Validation of the PROMIS tool for ASD
  2. Establish a core set of PROMs for best practice guidelines for ASD
  3. Evaluate patient reported outcome variance for ASD according to SRS-Schwab spine deformity type including variance in baseline PROM domains impacted and variance in improvement in PROM domains
  4. Evaluate ASD outcomes compared to population norms and investigate/develop appropriate measures of clinically significant improvement
* Evaluate clinical outcomes stratifying by patient chronological and physiological age
* Evaluate measures to quantify patient physiological age including patient frailty for ASD and validate a frailty measurement system for ASD
* Evaluate the role of functional tests in patient's baseline frailty assessment including hand manometer and Edmonton Frail Scale. See appendix, pages 17 & 18 for details.
* Evaluate the contribution of patient frailty to patient outcomes, complications, cost of care, disability, and complications
* Evaluate if patient frailty is a static measure or if frailty is a dynamic measure that can be improved through "pre-habilitation" and if the according associations with reductions in frailty correlate with reductions of cost, complications, and improvement in outcomes
* Evaluate cost variance for ASD surgery according to patient, institution, and geographical region and evaluate the cost effectiveness of surgical intervention for ASD
* Evaluate incidence of and risk factors for mental health (MH) compromise among ASD patients and establish best practice guidelines for assessing MH for ASD patients
* Evaluate the association of MH with surgical complications, outcomes, hospital length of stay and cost for ASD surgery
* Evaluate the association of social health surgical complications, outcomes, hospital length of stay and cost for ASD surgery and risk factors for routine (home) discharge vs. skilled nursing facility (SNF)/rehabilitation facility
* Broaden the evaluation of the surgically treated ASD patient to maximize evaluation of the entirety of the episode of care to include steps that can be taken prior to surgery including "prehabilitation," pain management, and MH care to improve treatment outcomes, reduce cost, reduce hospital length of stay, reduce non-routing discharge and reduce early and late complications
* Establish a core set of standard work guidelines to clinically and radiographically evaluate and treat ASD patients and evaluate the utility of standard work to improve outcomes for ASD and formulate best practice guidelines for surgical treatment of ASD
* Develop predictive analytic algorithms to risk stratify for best/worst outcomes, complications, sentinel events, and economic loss for ASD surgery
* Evaluate the prevalence and incidence of sacroiliac pain before/after complex adult spinal deformity surgery.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age at the time of treatment
2. EOS full body or standing 36" AP & Lateral images of entire spine
3. Posterior spine fusion with pedicle screw fixation construct of 5 or more levels
4. Pedicle screw fixation to be supplemented proximally with NuVasive VersaTie system
5. Upper instrumented vertebra (UIV) terminating at a newly instrumented level
6. Lowest instrumented vertebra (LIV) sacrum/pelvis
7. Surgery scheduled to take place in the next 6 months

Exclusion Criteria:

1. Active spine tumor or infection
2. Deformity due to acute trauma
3. Prisoners
4. Women who are pregnant
5. Patient is unwilling or unable to complete questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multicenter, prospective, observational, study evaluating the safety and performance of the VersaTie System by comparing adult patients receiving minimum 5 level posterior spinal fusion with pedicle screw fixation supplemented at the proximal aspect of the construct with the VersaTie System
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2021-07-09 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Scoliosis Research Society (SRS) 22r | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Scoliosis specific patient reported outcome
Oswestry | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Spine specific patient reported outcome
Veterans RAND 12 Item Health Survey (VR-12) | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Patient reported outcome
Patient-Reported Outcome Measurement Information System (PROMIS) - Anxiety | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Patient reported outcome
Patient-Reported Outcome Measurement Information System (PROMIS) - Depression | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Patient reported outcome
Patient-Reported Outcome Measurement Information System (PROMIS) - Pain Interference | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Patient reported outcome
Patient-Reported Outcome Measurement Information System (PROMIS) - Physical Function | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Patient reported outcome
Patient-Reported Outcome Measurement Information System (PROMIS) - Social Satisfaction | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Patient reported outcome
Patient-Reported Outcome Measurement Information System (PROMIS) - Social Role | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Patient reported outcome
Visual Analog Scale - Back Pain | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Self-reported back pain on scale of 0 (No pain) to 10 (severe pain)
Visual Analog Scale - Leg Pain | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Self-reported leg pain on scale of 0 (No pain) to 10 (severe pain)

SECONDARY OUTCOMES:
Edmonton Frail Scale | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Evaluate frailty on scale of 0 to 17 where higher scores mean more frail
Canadian Study of Health and Aging (CSHA) | Change from Preop to 3 months and 1, 2, 5 & 10 year follow-up
  Frailty scale of 1 to 9; higher scores mean more frail
Adverse Events | 3 months and 1, 2, 5 & 10 year post treatment
  Occurrence of Adverse events meeting reporting criteria and their relationship to intervention throughout the study
  [Time Frame: 3 months and 1, 2, 5 & 10 year post treatment]

CONTACTS AND LOCATIONS:
Overall Officials: Shay Bess, MD, Principal Investigator — Presbyterian/St Luke's Medical Center; Jeffrey Mullin, MD, Principal Investigator — University at Buffalo, Department of Neurosurgery; Christopher Shaffrey, MD, Principal Investigator — Duke University Medical Center, Section of Spine Surgery; Justin Smith, MD, Principal Investigator — University of Virginia Medical Center, Department of Neurosurgery
Locations (9):
- United States (9):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Shiley Center for Orthopaedic Research and Education at Scripps Clinic, La Jolla, California
  - University of California - San Francisco, San Francisco, California
  - Presbyterian/St. Luke's Medical Center, Denver, Colorado
  - Louisiana Spine Institute, Shreveport, Louisiana
  - University at Buffalo, Department of Neurosurgery, Buffalo, New York
  - New York University, Department of Orthopedic Surgery, New York, New York
  - Duke University Health System, Durham, North Carolina
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No